CLINICAL TRIAL: NCT05983835
Title: Combined Segmentectomy Versus Lobectomy for Stage IA Lung Adenocarcinoma With Ground-glass Component of Prospective, Randomized, Controlled Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Union-01
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2022-10

CONDITIONS: IA Lung Adenocarcinoma; Combined Segmentectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined segmentectomy (Experimental)
  Interventions: Procedure: Patients receive subsegmentectomy
- lobectomy (Placebo Comparator)
  Interventions: Procedure: Patients receive subsegmentectomy

INTERVENTIONS:
Procedure: Patients receive subsegmentectomy — Patients receive lobectomy

SUMMARY:
This project intends to include stage IA lung adenocarcinoma patients with CT imaging grboreal lesions; compare the results of lobectomy vs combined subsegmentectomy, and compare perioperative complications, differences in lung function and long-term outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age: 20-80 years, (2)suspected non-small-cell lung carcinoma, mixed nodules with GGO in the middle and peripheral lung fields, (3) clinical stage (UICC Stage 8) , Stage IA (T1a-cN0M0) , (4) multiple GGO was considered to be multiple primary lung cancer, but the largest diameter of GGO was less than 3 cm, the largest diameter of compactness was less than 2 cm, the largest diameter of GGO was less than 3 cm, the largest diameter of compactness was less than 2 cm, the largest diameter of GGO was less than 3 cm, the largest diameter of compactness was less than 2 cm (5) without any induction therapy; (6) PS score of 0-1, without severe complications, and functional status tolerant to minimally invasive lobectomy.

  (7) FEV1≥1L was assessed by pulmonary function test and was greater than 50% of the predicted value, (8) no hilar and mediastinal lymph node metastasis and no distant metastasis were found in the preoperative clinical evaluation, (9) voluntary participation and informed consent were obtained;

Exclusion Criteria:

* (1) pure dense nodules without GGO, or pure GGO ≤0.5 cm with GGO;(2) the lesion was located in 1/3 of the lung field, and combined segmental resection may not meet the requirement of resection margin (3) multiple GGO considered multiple primary lung cancer with the largest diameter ≥1cm, dense component ≥0.5 cm and a second primary lesion that may require surgical treatment in the next 5 years (4) high risk patients with severe other organ diseases, (5) history of other malignant tumors within 5 years, (6) history of ipsilateral thoracic surgery. (7) the lesion was located in the middle lobe of the right lung, (8) in pregnant or lactating women, (9) with severe mental disorders, (10) with a history of unstable angina or myocardial infarction within 6 months, and severe stenosis of the major branches of the coronary artery; (11) a history of cerebral infarction or cerebral hemorrhage within 6 months, (12) a history of continuous systemic corticosteroid therapy within 1 month, and (13) according to the judgment of the investigators, the patients were not suitable to be included in the trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 2 years
  This is the time from the time of surgery until the patient's tumor recurred, metastasized, or died

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, China